CLINICAL TRIAL: NCT04202133
Title: A Randomized Controlled Trial Examining the Neurocognitive Benefits of a Nationally Available Weight Management Program
Brief Title: Neurocognitive Benefits of a Weight Management Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 834404
Record Dates: First submitted 2019-12-03; First posted 2019-12-17 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Overweight and Obesity
Keywords: obesity; weight loss; neuroimaging; fMRI; behavioral obesity treatment
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WW (formerly Weight Watchers) (Experimental): 16-weeks of the group-based WW program
  Interventions: Behavioral: WW (formerly Weight Watchers)
- Waitlist Control (Other): 16-weeks on waitlist then participants will be provided with 16-weeks of the group-based WW program
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: WW (formerly Weight Watchers) — The WW intervention will consist of weekly group workshops for 16 weeks with WW Coaches and Guides.
  Arms: WW (formerly Weight Watchers)
Behavioral: Waitlist — The waitlist group will have a 16-week waitlist period. After the waitlist period, they will be offered the WW intervention
  Arms: Waitlist Control

SUMMARY:
This study will assess whether weight loss induced through diet and physical activity can change neural responses to high- and low-calorie food images. In addition, it will evaluate whether weight loss can improve neural function when performing the N-back task, a measure of working memory. Findings will address notable gaps in the literature by testing whether a scalable weight loss intervention can help protect and improve neurocognitive functioning and brain health in individuals with obesity. This study will also provide important information about the effects of weight loss on neuroplasticity in brain regions crucial for memory and cognitive functioning, which will help to inform future interventions aimed at promoting brain health.

DETAILED DESCRIPTION:
The purpose of the present study is to conduct a randomized controlled trial (RCT) to assess the effects of a commercially available weight loss program (WW; formerly Weight Watchers) on neural response to food cues and memory tasks, as well as on structural brain morphology. Participants with obesity will be randomized to either 16 weeks of an in-person, group-based WW program (n=30) or a wait-list control (WLC; n=30). Both groups will have structural and blood oxygen level-dependent (BOLD) functional magnetic resonance imaging (fMRI) scans at baseline and after the 16-week intervention. Participants will complete the following fMRI tasks: 1) structural scan; 2) food cue task to measure reactivity to high and low-calorie food images and 3) N-back task to measure working memory (i.e., the ability to temporarily hold information available for processing). In addition, participants will complete self-report and behavioral measures of eating behaviors, appetite, physical activity, mood, quality of life, attention and memory at baseline, and weeks 8 and 16.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60 years
* Female
* BMI>30 kg/m2
* Eligible female patients will be:

  * Non-pregnant
  * Non-lactating
  * Surgically sterile or postmenopausal, or they will agree to continue to use an accepted method of birth control during the study. Acceptable methods of birth control are: hormonal contraceptives; double barrier method (condom with spermicide or diaphragm with spermicide); intrauterine device; surgical sterility; abstinence; and/or postmenopausal status (defined as at least 2 years without menses).
* Participants must:

  * Understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent

Exclusion Criteria:

* Weight>158.8 kg (350 lbs, due to scanner weight restrictions)
* Serious medical risk such as type 1 or 2 diabetes, cancer, or recent cardiac event (e.g., heart attack, angioplasty)
* Untreated thyroid disease or any changes (type or dose) in thyroid medication in the last 6 months
* Current psychiatric disorder that significantly interferes with daily living
* Active suicidal ideation
* Current substance use disorder (current or in remission < 1 year)
* Presence or history of orthopedic circumstances, metallic inserts, pacemaker, claustrophobia, or other conditions that may interfere with magnetic resonance imaging
* Participation in a structured weight loss program in the prior 6 months
* WW member within the past 12 months
* Use of medications known to induce significant weight loss/gain, including chronic use of oral steroids in the past 3 months
* Psychiatric hospitalization within the past 6 months
* Loss of >10 lbs of body weight within the past 3 months
* History or plans for bariatric surgery
* Visual, auditory, or other impairment affecting task performance
* Epilepsy
* Neurological trauma (e.g., concussion)
* Inability to attend treatment and/or assessment visits
* Participant from same household
* Adherence to specialized diet regimes, such as vegetarian, macrobiotic
* Lack of capacity to provide informed consent
* Inability to walk 5 blocks comfortably or engage in some other form of aerobic activity (e.g., swimming)
* Any serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safety or successful participation in the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 61 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariana M. Chao, PhD, CRNP, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chao AM, Wadden TA, Cao W, Zhou Y, Maldonado D, Cardel MI, Foster GD, Loughead J. Randomized Controlled Trial of Effects of Behavioral Weight Loss Treatment on Food Cue Reactivity. Nurs Res. 2024 Mar-Apr 01;73(2):91-100. doi: 10.1097/NNR.0000000000000702. Epub 2023 Oct 31. PMID 37916843
- [Derived] Chao AM, Zhou Y, Erus G, Davatzikos C, Cardel MI, Foster GD, Wadden TA. A randomized controlled trial examining the effects of behavioral weight loss treatment on hippocampal volume and neurocognition. Physiol Behav. 2023 Aug 1;267:114228. doi: 10.1016/j.physbeh.2023.114228. Epub 2023 May 6. PMID 37156318

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Started | 31 | 30
Completed | 30 | 26
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8.7) | 40.1 (11.1) | 41.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 15 | 31
  White | 13 | 13 | 26
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level-dependent (BOLD) Response to High-calorie Foods Cues Minus Neutral Objects in Left Anterior Cingulate Cortex
Description: Changes in BOLD fMRI response to high-calorie food images
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: percent BOLD signal change
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 29 | 22
percent BOLD signal change | -0.05 (0.05) | -0.16 (0.06)

2. Primary Outcome: Reward-based Eating
Description: Changes in scores on the Reward-Based Eating Drive Scale; range of 0-52; higher scores indicate higher reward-related eating
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 30 | 26
units on a scale | -3.9 (1.4) | -0.7 (1.5)

3. Primary Outcome: Food Cravings- Trait (Lack of Control Over Eating)
Description: Changes in scores on the Food Cravings Questionnaire- Trait (lack of control over eating), range=6-36, higher scores indicate greater cravings
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 31 | 30
score on a scale | -2.7 (0.8) | -0.1 (0.9)

4. Primary Outcome: Food Preference
Description: Changes in scores on the Leeds Food Preference Questionnaire
Time Frame: Change from baseline to 16 weeks
Population: Data not analyzed due to technical error with coding of the task that resulted in the data being unusable
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Eating Behaviors
Description: Changes in scores on the Eating Behaviors Questionnaire (liking for high-calorie foods); visual analog scores ranging from 0-100 with higher scores indicating a worse outcome
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 31 | 30
units on a scale | -3.2 (2.1) | 1.0 (2.3)

6. Primary Outcome: Hippocampal Volume
Description: Change in hippocampal volume
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 29 | 22
mm^3 | -84.9 (154.8) | 42.8 (172.9)

7. Primary Outcome: BOLD fMRI Response to the N-back Task
Description: Changes in BOLD fMRI response to the N-back task
Time Frame: Change from baseline to 16 weeks
Population: Data not analyzed due to technical error due to coding in N-bask task in E-Prime that resulted in the data being unusable
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Eating Behaviors (Low-calorie Foods)
Description: Changes in scores on the Eating Behaviors Questionnaire (liking for low-calorie foods); visual analog scores ranging from 0-100 with higher scores indicating a better outcome
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 31 | 30
units on a scale | 0.7 (2.3) | -0.8 (2.3)

9. Secondary Outcome: N-back Behavioral Performance
Description: Change in reaction time (seconds) on the N-back task
Time Frame: Change from baseline to 16 weeks
Population: as for outcome 7
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percent Weight
Description: Percent weight change
Time Frame: Change from baseline to 16 weeks
Measure: Mean (Standard Error); unit: percentage of initial weight loss
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 31 | 30
percentage of initial weight loss | -4.7 (4.9) | 0.2 (3.5)

11. Secondary Outcome: Eating Behavior
Description: Changes in eating behavior as measured by the Eating Inventory (Cognitive restraint, disinhibited eating, and hunger subscales, summed scores, higher values indicate greater restraint/disinhibition/hunger). The cognitive restraint scale includes 21 items (range 0-21). Higher scores demonstrate more awareness of one's eating and success in restricting dietary intake for weight control. The disinhibited eating scale includes 16 items (range 0-16). Higher scores signify more overeating tendencies. The hunger scale has 14 items and higher scores indicate more perceived hunger (range 0-14). Subscales were analyzed separately.
Time Frame: Change from baseline to 16 weeks
Population: Intention to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 30 | 26
score on a scale
  Cognitive restraint | 3.5 (0.6) | 0.3 (0.7)
  Hunger | -0.9 (0.4) | -0.7 (0.5)
  Disinhibition | -1.5 (0.4) | -0.4 (0.5)

12. Secondary Outcome: Power of Food
Description: Changes in eating behavior as measured by the Power of Food Scale; higher scores indicate greater hedonic hunger. Range of scores is 1-5
Time Frame: Change from baseline to 16 weeks
Population: Intention to treat
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
Number analyzed (Participants) | 30 | 26
score on a scale | -0.4 (0.6) | -0.1 (0.7)

ADVERSE EVENTS:
Time Frame: Baseline and follow-up (16 weeks)
Arm/Group | WW (Formerly Weight Watchers) | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT04202133/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT04202133/SAP_001.pdf